CLINICAL TRIAL: NCT01632839
Title: Psychometric Validation of a French Version of the PISQ-R and a New Questionnaire About Sexuality: Tools for Evaluating Sexuality in Patients With From Urinary Incontinence or Pelvic Organ Prolapse
Brief Title: Psychometric Validation of a French Version of the PISQ-R and a New Questionnaire About Sexuality
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2011/BF-03; 2012-A00303-40 (Other: ANSM)
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2017-07

CONDITIONS: Sexuality; Pelvic Organ Prolapse; Urinary Incontinence; Fecal Incontinence
Keywords: PISQ-R; new sexuality questionnaire
MeSH Terms: conditions — Sexuality; Pelvic Organ Prolapse; Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Vaginal surgery +prothesis +sexuality: The 50 patients included in this group will have undergone vaginal surgery for pelvic organ prolapse with placement of a prothesis; these patients are sexually active.
- Vaginal surgery +prothesis -sexuality: The 25 patients included in this group will have undergone vaginal surgery for pelvic organ prolapse with placement of a prothesis; these patients are NOT sexually active.
- Vaginal surgery -prothesis + sexuality: The 50 patients included in this group will have undergone vaginal surgery for pelvic organ prolapse WITHOUT placement of a prothesis; these patients are sexually active.
- Vaginal surgery -prothesis -sexuality: The 25 patients included in this group will have undergone vaginal surgery for pelvic organ prolapse WITHOUT placement of a prothesis; these patients are NOT sexually active.
- Abdominal surgery +sexuality: The 50 patients included in this group will have undergone abdominal surgery for pelvic organ prolapse; these patients are sexually active.
- Abdominal surgery -sexuality: The 25 patients included in this group will have undergone abdominal surgery for pelvic organ prolapse; these patients are NOT sexually active.
- Urinary incontinence surgery + sexuality: The 50 patients included in this group will have surgery for urinary incontinence; these patients are sexually active.
- Urinary incontinence surgery - sexuality: The 25 patients included in this group will have surgery for urinary incontinence; these patients are NOT sexually active.

SUMMARY:
The primary objective of this study is the psychometric validation of two questionnaires (PISQ-R and a new questionnaire on sexuality) as compared to a non specific questionnaire on female sexual function (FSFI).

ELIGIBILITY:
Inclusion Criteria:

* Patient is not pregnant
* Patient can read and understand French
* The patient must have given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has genital prolapse and/or urinary incontinence and/or anal incontinence, and have undergone surgery

Exclusion Criteria:

* The patient is under judicial protection
* The patient does not understand french
* Patient has vulvodynia
* Patient has painful bladder syndrome
* The patient has had chronic pelvic pain for longer than 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing vaginal, abdominal or urinary incontinence surgery.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2013-01-18 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
PISQ-R questionnaire | 12 months + 1 week

SECONDARY OUTCOMES:
PISQ-R questionnaire | baseline; day 0
PISQ-R questionnaire | 6 months
PISQ-R questionnaire | 12 months
New sexuality questionnaire | baseline; day 0
New sexuality questionnaire | 6 months
New sexuality questionnaire | 12 months
New sexuality questionnaire | 12 months + 1 week
PFDI questionnaire | baseline; day 0
PFDI questionnaire | 6 months
PFDI questionnaire | 12 months
ICI-Q questionnaire | baseline; day 0
ICI-Q questionnaire | 6 months
ICI-Q questionnaire | 12 months
FSFI questionnaire | baseline; day 0
FSFI questionnaire | 6 months
FSFI questionnaire | 12 months
PGI-I questionnaire | baseline; day 0
PGI-I questionnaire | 6 months
PGI-I questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Renaud de Tayrac, MD PhD, Study Director — Centre Hospitalier Universitaire de Nîmes; Brigitte Fatton, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (14):
- France (14):
  - APHP - Hôpital Antoine Beclere, Clamart
  - CHU de Clermont Ferrand - Hôpital Estaing, Clermont-Ferrand
  - G.C.S. Flandre Maritime - site Polyclinique de Grande-Synthe, Grande-Synthe
  - CH de la Rochelle, La Rochelle
  - APHP - Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - CHRU de Lille - Hôpital Jeanne de Flandre, Lille
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Groupe Hospitalier Dioconesses - Site Reuilly, Paris
  - APHP - Hôpital Bichat - Claude Bernard, Paris
  - CHU de Poitiers, Poitiers
  - CH de la Région d'Annecy, Pringy
  - CH de Poissy - Saint-Germain-en-Laye, Saint-Germain-en-Laye
  - CHRU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes

REFERENCES:
- [Result] Fatton B, Hermieu JF, Lucot JP, Debodinance P, Cour F, Alonso S, de Tayrac R. French validation of the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire-IUGA revised (PISQ-IR). Int Urogynecol J. 2021 Dec;32(12):3183-3198. doi: 10.1007/s00192-020-04625-6. Epub 2021 Jan 5. PMID 33399902